CLINICAL TRIAL: NCT02985697
Title: Safety and Efficacy of Intranasal Dexmedetomidine as a Sedative in Pediatric Dentistry: a Randomized, Double-blind Clinical Study
Brief Title: Safety and Efficacy of Intranasal Dexmedetomidine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bon Secours Pediatric Dental Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8001
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Safety and Efficacy of Intranasal Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IN DEX (Experimental): Group IN DEX will receive a placebo dose of flavored water followed by 3 mcg/kg intranasal dexmedetomidine in conjunction with 50/50 nitrous oxide/oxygen at a calculated flow rate. If adequate sedation is not obtained within 60 minutes of drug administration, the sedation will be considered a failure and the procedure will be terminated and rescheduled for completion of care using deep sedation or general anesthesia, in keeping with normal office policy. Second doses of intranasal dexmedetomidine or placebo will not be given.
  Interventions: Drug: Dexmedetomidine; Drug: Nitrous Oxide
- MIDDEX (Experimental): Group MIDDEX will receive 3 mcg/kg intranasal dexmedetomidine and 0.5 mg/kg oral midazolam and 100% oxygen at a calculated flow rate (oxygen administration to function as placebo for nitrous oxide). If adequate sedation is not obtained within 60 minutes of drug administration, the sedation will be considered a failure and the procedure will be terminated and rescheduled for completion of care using deep sedation or general anesthesia, in keeping with normal office policy. Second doses of intranasal dexmedetomidine or oral midazolam will not be given.
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam Hydrochloride
- NOMIDDEX (Experimental): Group NOMIDDEX will receive 3 mcg/kg intranasal dexmedetomidine, 0.5 mg/kg oral midazolam, and 50/50 nitrous oxide/oxygen at a calculated flow rate. If adequate sedation is not obtained within 60 minutes of drug administration, the sedation will be considered a failure and the procedure will be terminated and rescheduled for completion of care using deep sedation or general anesthesia, in keeping with normal office policy. Second doses of intranasal dexmedetomidine or oral midazolam will not be given.
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam Hydrochloride; Drug: Nitrous Oxide
- CTRL (Active Comparator): The control group, Group CTRL, will receive a placebo dose of normal saline and 0.5 mg/kg oral midazolam and 50/50 nitrous oxide/oxygen at a calculated flow rate. Midazolam was chosen as the control due to its well documented history of use in pediatric procedural sedations. If adequate sedation is not obtained within 60 minutes of drug administration, the sedation will be considered a failure and the procedure will be terminated and rescheduled for completion of care using deep sedation or general anesthesia, in keeping with normal office policy. Second doses of intranasal dexmedetomidine or oral midazolam will not be given.
  Interventions: Drug: Midazolam Hydrochloride; Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Dexmedetomidine — The intervention being tested is intranasal dexmedetomidine
  Other Names: Precedex; Dexdor; Dexdomitor; Sileo
  Arms: IN DEX; MIDDEX; NOMIDDEX
Drug: Midazolam Hydrochloride — Oral midazolam is being used as the Active Comparator. It will also be used in conjunction with IN dexmedetomidine in some experimental groups.
  Other Names: Versed
  Arms: CTRL; MIDDEX; NOMIDDEX
Drug: Nitrous Oxide — Nitrous oxide to be administered in conjunction with other interventions, per study design.
  Arms: CTRL; IN DEX; NOMIDDEX

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of intranasal dexmedetomidine when used in combination with oral midazolam and/or nitrous oxide for moderate sedation during pediatric outpatient dental procedures.

DETAILED DESCRIPTION:
The study will be organized as a prospective, randomized, double-blind trial in which children who meet the study criteria are randomly separated into three test groups (IN DEX, MIDDEX, and NOMIDDEX) and one control group (CTRL). Patients will be scheduled to complete one quadrant of dental care per sedation. Dental procedures to be performed include composite restorations, sealants, stainless steel crowns, pulp therapy, and extractions, with the exact number and type dependant on each patient's individual treatment plan.

Group IN DEX will receive a placebo dose of flavored water followed by 3 mcg/kg intranasal dexmedetomidine in conjunction with 50/50 nitrous oxide/oxygen at a calculated flow rate. If adequate sedation is not obtained within 60 minutes of drug administration, the sedation will be considered a failure and the procedure will be terminated and rescheduled for completion of care using deep sedation or general anesthesia, in keeping with normal office policy. Second doses of intranasal dexmedetomidine or placebo will not be given.

Group MIDDEX will receive 3 mcg/kg intranasal dexmedetomidine and 0.5 mg/kg oral midazolam and 100% oxygen at a calculated flow rate (oxygen administration to function as placebo for nitrous oxide). If adequate sedation is not obtained within 60 minutes of drug administration, the sedation will be considered a failure and the procedure will be terminated and rescheduled for completion of care using deep sedation or general anesthesia, in keeping with normal office policy. Second doses of intranasal dexmedetomidine or oral midazolam will not be given.

Group NOMIDDEX will receive 3 mcg/kg intranasal dexmedetomidine, 0.5 mg/kg oral midazolam, and 50/50 nitrous oxide/oxygen at a calculated flow rate. If adequate sedation is not obtained within 60 minutes of drug administration, the sedation will be considered a failure and the procedure will be terminated and rescheduled for completion of care using deep sedation or general anesthesia, in keeping with normal office policy. Second doses of intranasal dexmedetomidine or oral midazolam will not be given.

The control group, Group CTRL, will receive a placebo dose of normal saline and 0.5 mg/kg oral midazolam and 50/50 nitrous oxide/oxygen at a calculated flow rate. Midazolam was chosen as the control due to its well documented history of use in pediatric procedural sedations. If adequate sedation is not obtained within 60 minutes of drug administration, the sedation will be considered a failure and the procedure will be terminated and rescheduled for completion of care using deep sedation or general anesthesia, in keeping with normal office policy. Second doses of intranasal dexmedetomidine or oral midazolam will not be given.

The initial flow rate of nitrous oxide/oxygen will be calculated by multiplying the patient's respiratory rate by their estimated tidal volume. Tidal volume is estimated at 10 ml/kg. The flow rate will then adjusted to the patient's pulmonary needs. At the conclusion of the procedure, all patients will be given 100% oxygen for at least 5 minutes and allowed to recover to stable vital signs, level of consciousness, motor function, and adequate hydration and pain control before discharge.

All intranasal drugs and placebos will be administered using the MAD300 Nasal Drug Delivery Device, manufactured by Wolfe Tory. Typical particle size delivered into the nare is 30-100 microns. The device is 1.65 inches in length, has a tip diameter of .17 inches, and an internal dead space of 0.07 ml. Dexmedetomidine will be drawn from the manufacturer's vial and administered non-diluted (200 mcg/ml). The medication will be administered nearly immediately (less than 1 minute from withdrawal from original vial). A maximum of 1ml will be administered per nare.

All nasal administration of drugs and placebos will occur approximately 30 minutes before scheduled procedure start time and all orally administration of drugs and placebos will occur approximately 15 minutes before scheduled procedure start time. Administration of all inhaled agents and placebos will begin approximately 5 minutes prior to scheduled procedure start time. This delay will allow for coincident onset of drug effects.

In accordance with Bon Secours policy and evidence based guidelines, vital signs of all patients will be monitored by a Bon Secours nurse from the time of drug administration until discharge. Pulse oximetry, heart rate, respiratory rate, and end tidal CO2 will be monitored continuously. Blood pressure will be measured via an appropriately sized arm cuff every 5 minutes, beginning 5 minutes prior to first drug or placebo administration and ending when the patient meets discharge criteria. The sedating dentist will be present in a supervisory role for the duration of the sedation and remain immediately available until the patient is discharged.

In accordance with Bon Secours policy, all patients will be required to have a history and physical completed by their primary care provider a maximum of 30 days prior to date of procedure. Patients are also required to observe hospital pre-operative fasting guidelines (NPO solids, milk, formula > 6 hours, breast milk > 4 hours, clear liquids > 2 hours). Topical and local anesthesia (2% lidocaine with 1:100,000 epinephrine) will be administered prior to operative procedures to facilitate pain control. Patient caregivers will be given appropriate post-operative instructions. Each patient will be followed up with a phone call the evening of the procedure and the next day to inquire about any complications and whether or not the child has returned to baseline activity.

Age, weight, gender, ASA status, dosages of all drugs used, monitoring provider, procedural times, adverse events, required interventions, and quality of sedation will be recorded. Apnea, desaturation, airway obstruction, bradycardia, hypotension, fever, and inability to complete the procedure will be considered minor adverse events. Major adverse events are defined as death, aspiration, cardiac arrest, unplanned hospital admission, and level-of-care increase.

If a patient has 3 consecutive blood pressure readings (taken at 5 minute intervals) that fall below the 5th percentile for age, the hypotension protocol will be initiated. The hypotension protocol consists of: (1) Placement of an IV. (2) Administration of 20 ml/kg of IV normal saline every 5 minutes (maximum of 60 ml/kg over 15 minutes) (3) Concentration of nitrous oxide will be reduced to 25%, if applicable and no additional sedative agents will be administered (4) If blood pressure improves with intervention and the patient remains adequately sedated, the scheduled dental procedures will be completed. (5) If intervention is unsuccessful and blood pressure does not improve, the procedure will be terminated and the patient will be transferred to the emergency room for level of care increase.

In the event that a patient experiences rage, agitation, or paradoxical excitation, they will be restrained using protective stabilization for their safety. Consent for protective stabilization will be obtained when consent for sedation and study participation is obtained.

Patient olfaction will be assessed preoperatively and postoperatively using standard anesthesia olfactory oils when possible (based on pt age and developmental status). Nasal mucosa will be examined preoperatively and postoperatively by the attending sedationist. Abnormalities will be referred to the patient's primary care provider.

Sedation quality and patient behavior will be evaluated using the University of Michigan sedation scale.

Safety will be assessed by analyzing adverse events. Efficacy will be assessed by analyzing the quality of sedation based on scoring from the University of Michigan Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 3 through 6 years of age.
2. Patients who are appropriate for in-office sedation for dental care.

Exclusion Criteria:

1. Patients younger than 3 or older than 6 years of age.
2. History of failed sedation.
3. BMI greater than 30.
4. Patients weighing less than 10 kgs.
5. Patients weighing more than 25 kgs.
6. Patients who are deemed unsuitable for sedation by a physician at their preoperative history and physical.
7. Patients who are deemed unsuitable for in-office sedation in accordance with Bon Secours policy (American Society of Anesthesiologists [ASA] Classification greater than II, Mallampati score greater than 2, Brodsky tonsil score greater than 2).
8. Patients with sleep apnea.
9. Patients with a history of an unfavorable reaction to DEX or clonidine.
10. Patients with pulmonary hypertension.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 1 year
  Apnea, desaturation, airway obstruction, bradycardia, hypotension, fever, and inability to complete the procedure will be considered minor adverse events. Major adverse events are defined as death, aspiration, cardiac arrest, unplanned hospital admission, and level-of-care increase. Required interventions to correct adverse events will also be recorded (such as IV fluids to improve hypotension).
Quality of Sedation | 1 year
  Sedation quality and patient behavior will be evaluated using the criteria from the University of Michigan sedation scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Bon Secours Pediatric Dental Associates, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol: DEXProtocol — https://drive.google.com/open?id=0BwBFaEmsvS0PYnlzVDUyMGREWFk — Protocol for the study; includes introduction, design, and references/citations.